CLINICAL TRIAL: NCT03346226
Title: Influence on Incidence of Postoperative Delirium by Various Sedatives in Elderly Patients With Hip Fracture Under Lumbar Anesthesia: A Randomized, Control and Multi-center Trial
Brief Title: How Different Sedatives Affect Hip Fracture Patient's Postoperative Delirium
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); The Second Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Nanchang University (Other); Qianfoshan Hospital (Other); Shanghai 6th People's Hospital (Other); Tang-Du Hospital (Other); Second Hospital of Shanxi Medical University (Other); The First Affiliated Hospital of Soochow University (Other); Shanghai Changzheng Hospital (Other); The Fuzhou No 2 Hospital (Other); Foshan Hospital of Traditional Chinese Medicine (Other); Beijing Jishuitan Hospital (Other)
Responsible Party: Principal Investigator, Guowei Tu, director of Anesthesiology Department, Principal Investigator, Clinical Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Postoperative Delirium
Record Dates: First submitted 2017-09-14; First posted 2017-11-17 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Delirium in Old Age
Keywords: Delirium Dexmedetomidine elderly
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Intervention Model Description: Dexmedetomidine group：dexmedetomidine is given to patients under spinal anesthesia until the end of surgery propofol group:Propofol is given to patients uunder spinal anesthesia until the end of surgery
Who Masked: Outcomes Assessor
Masking Description: the intervention is happend in the operation，the outcome assessment is going after the operation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine Hydrochloride (Experimental): Dex Group: 0.5 μg/kg of Dex is given 10 minutes before operation through injection pump during 15 minutes. After the operation starts, the initial pumping ratio of Dex is 0.5ug/kg/h and adjusted under BIS surveillance to keep BIS between 70-80 until 30 minutes before the end of surgery. Meanwhile, OAA/S grade is evaluated every 15 minutes to maintain OAA/S at grade 4. If discrepancy occurs, OAA/S prevails.
  Interventions: Drug: Dexmedetomidine Hydrochloride
- Propofol (Active Comparator): Prop Group: Propofol is given with an initial ratio of 2-10mg/kg/h, when the operation starts. Under BIS surveillance, dripping rate is adjusted to keep BIS between 70-80 until 5 minutes before the end of surgery. Meanwhile, OAA/S grade is evaluated every 15 minutes to maintain OAA/S at grade 4. If discrepancy occurs, OAA/S prevails.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Dexmedetomidine is given to patients during spinal anesthesia at the dose of 0.5 μg/kg，adjusted the dose to keep BIS between 70-80 until 30 minutes before the end of surgery
  Other Names: brand name ：YiSi
  Arms: Dexmedetomidine Hydrochloride
Drug: Propofol — Propofol is given with an initial ratio of 2-10mg/kg/h, when the operation starts，adjust the propofol's dose to keep BIS between 70-80 before the end of surgery
  Other Names: Brand name：Diprivan or other brands of propofol
  Arms: Propofol

SUMMARY:
the hypothesis is that Dexmedetomidine seems to decrease incidence of post-operative delirium . one possible mechanism is that Dex have a minor influence on cognition, since it has no effect on GABA receptor，another is that Dex could induce a sleep similar to natural sleep, thereby decreasing sleep deprivation and circadian rhythm disorder in post-operative patients.

In this study , investigators devise the two different sedatives(Dexmedetomidine and Propofol)'influence on postoperative delirium in hip fracture elderly participants under spinal anesthesia

DETAILED DESCRIPTION:
With a complex etiology, delirium is usually caused by various peri-operative stimuli on basis of predisposing factors, including senility, hypoxia and hypotension, pain, drug (such as pethidine, benzodiazepine, anticholinergic, and drug withdrawal), complications prior to surgery, post-operative sleep disorder. As for the mechanism of delirium, the commonly accepted hypothesis includes the decreased central cholinergic neurons function and the inflammation of central nervous system. Most of the hip fracture patients are senile, suffering generally from many complications with exposure to many drugs, and poor in nutritional status with decreased cognitive function even before the surgery in some of them, all of which are risk factors for post-operative delirium. Systematic review suggests that incidence of POD in patients undergoing elective hip arthroplasty is up to 4-53.3%. It is of great importance, therefore, to explore the effective approaches to lower POD incidence in senile patients with operation on hip fracture.

Dexmedetomidine Hydrochloride is a novel highly-selective α2 adrenergic receptor agonist, and its selectivity to α2 receptor is 8 times of that of clonidine. It has multiple functions including sedation, anti-anxiety, hypnosis, analgesia and sympathetic blockade, with a wide application prospect for peri-operative patients. Researches suggest that Dex applied peri-operatively may stabilize blood pressure and heart rate, control intra-operative stress, and decrease post-operative side reactions such as nausea, vomiting, restlessness, delirium and chills. Moreover, advantages of Dex also include analgesia and reduction of opioid usage. Clinical pharmacological characteristics of Dex suggest its possible function to decrease post-operative delirium. Meanwhile, Dex seems to have a minor influence on cognition, since it has no effect on GABA receptor.

Another important feature of it is that Dex induces a sleep similar to natural sleep, thereby decreasing sleep deprivation and circadian rhythm disorder in post-operative patients, and decreasing incidence of post-operative delirium. Researches evaluating the capability of Dex to decrease delirium incidence are focused on ICU sedation post to operation. Riker et al compared the sedative effect between Dex and midazolam in patients with severe mechanical ventilation, revealing a lower delirium incidence in Dex than in midazolam (54.0% vs 76.6%) in patients maintained with the same depth of sedation. Systematic review concludes that Dex in effective to prevent and treat post-operative delirium in ICU patients.

In this study ,the investigators devise the two different sedatives (Dexmedetomidine and Propofol)'influence on postoperative delirium in hip fracture elderly participants under spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

1. Acquisition of informed consent,
2. Patients with hip fracture surgery under lumbar anesthesia,
3. Grade II to III based on American Society of Anesthesiologists ASA classification,
4. Age ≥65 and ≤90 years old.

Exclusion Criteria:

1. History of psychiatric disease or a disease needing long-term exposure to psychotropic drugs (dementia, schizophrenia), or history of alcoholic abuse.
2. More than 8 errors in preoperative Simplified Psychology and Mental Status Questionnaire (SPMSQ) , and diagnosed as severe cognitive impairment.
3. CAM positive diagnosed preoperatively.
4. Any cerebrovascular accident occurring within 3 months, such as cerebral stroke or transient ischemic attack (TIA).
5. Systolic pressure < 90mmHg and diastolic pressure < 60mm Hg at the preoperative follow up or HR< 50/minute.
6. History of heat failure or EF<30% as shown by ultrasound cardiogram; degree 2 type 2 and degree 3 atrioventricular block. History of active heart disease (such as acute cardiac infarction, unstable angina pectoris)
7. Severe abnormality in hepatic or renal function (severe abnormality in liver function: more than 2-times increase than upper normal limit in any one of the markers including ALT,, conjugated bilirubin, AST, ALP, total bilirubin; severe abnormality in renal function; Cr clearance<30ml/min), Scr>443μmol/L.
8. Diabetes patients with severe complications of diabetes (Diabetic ketoacidosis, hyperosmolar coma, various infections, macrovascular diseases, and diabetic nephropathy)
9. Patients with severe infection.
10. Postoperative PaO2<60mmHg or SpO2<92%.
11. Participation in clinical trials of other drugs within past 30 days.
12. Disturbed verbal communication, and unable to accomplish the test on cognition.
13. Patients with prosthesis fracture or restoration; hip fracture but complicated with severe trauma in other sites.
14. Being allergic to investigational drug or having contradiction of lumbar anesthesia.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
occurrence of postoperative delirium in postoperative 72 hours | patient enrolled will be evaluated at 9Am and 3Pm during post-operative day 1-3 (POD1-3).At any time point above，delirium is detected，then the patient will be diagnosed as postoperative delirium. All patients enrolled is Non-delirium before surgery。
  Evaluation of delirium is performed by trained investigational assistant who does not know the randomization of patients. Follow up is carried out before operation and at 9Am and 3Pm during post-operative day 1-3 (POD1-3). During follow up, RASS (Richmond Agitation-Sedation Scale, RASS) is used firstly to evaluate sedation of the patients, and for those with ARSS >-4 (-3～+4), the Confusion Assessment Method (CAM) is adopted for evaluation. A case consistent with delirium standard at any time point during follow up is determined to be delirium positive. Diagnosis should be confirmed for a CAM-positive patient by a psychological expert based on DSM-V standard

SECONDARY OUTCOMES:
Consumption of analgesic | record the data of comsumption of analgeisic at 48 hours after operation
  the patients will receive patient-controlled intravenous analgesia，record the consumption of intravenous analgesia in the 48 postoperative hours
Times of intra-operative occurrence of hypotension, bradycardia, hypertension and tachycardia that need treatment. | during the operation
  assess the adverse effect of anaesthetic
Score of quality of post-operative sleeping | quality of sleeping will be assessed at 9Am during post-operative day 1-3
  Score of sleeping quality is evaluated based on the some questions during follow up
Hospital stay | record the days of hospital stay at the 30 days after surgery
  the duration from the day of operation to the date meeting discharge criteria as determined by doctor in charge
Post-operative complications besides delirium | observe and evaluate complications at the 30 days after surgery
  complications besides delirium ，such as vomiting，nausea，hypotention，hypertention，bradycardia
Mortality up to day 30 post to operation | the data will be collected after 30 days of operation
  Data for 30-day survival is collected through telephone follow up by the assistant.
pain score | Pain score will be evaluated at time point of operation, 1，6，24, 48 hours after operation, using NRS score
  describe severity of the pain the patient feel using Numerical Rating Scale （NRS）

CONTACTS AND LOCATIONS:
Overall Officials: Xue ZhangGang, doctor, Principal Investigator — Anesthesiology Department of Shanghai Zhongshan Hospital